CLINICAL TRIAL: NCT00434551
Title: Evaluation of Capsule Endoscopy in Patients With Suspected Small Bowel Crohn's Disease
Brief Title: MACCS: Multicenter Australian CE in Patients With Suspected Crohn's Disease Study
Acronym: MACCS
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Corporate Director Clinical Affairs, Given Imaging Ltd.
Other Study IDs: MA-36
Record Dates: First submitted 2007-02-11; First posted 2007-02-13 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2007-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: small bowel Crohn's disease; capsule endoscopy; PillCam SB; Patients with suspected small bowel Crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with suspected Crohn's disease

SUMMARY:
This is a prospective study aimed to validate the ability of capsule endoscopy to accurately diagnose small bowel Crohn's disease in symptomatic patients who have a non-diagnostic standard workup. Patients will be randomized to undergo capsule endoscopy either one week or five weeks after enrolment. Patients will be followed up for up to 3 months after capsule endoscopy.

DETAILED DESCRIPTION:
In the past few years, capsule endoscopy has sparked renewed interest in the investigation of small bowel Crohn's disease. A PillCam™SB capsule (Given Imaging Ltd, Yoqneam, Israel) is an ingestible, disposable video camera that transmits high quality images of the small intestinal mucosa. This enables the small intestine to be readily accessible to physicians investigating for the presence of small bowel disorders such as Crohn's disease. It has been demonstrated that capsule endoscopy identifies Crohn's disease when other methods are not helpful. Diagnostic yields of 70% have been reported in small series of studies performed in suspected small bowel Crohn's disease.

This study is designed to determine the accuracy and clinical impact of Capsule Endoscopy in detecting suspected small Bowel Crohn's Disease whose initial evaluation was non-diagnostic. It will also serve to better understand the impact of capsule endoscopy on the natural history of the disorder.

Patients will be randomized to undergo capsule endoscopy either one week or five weeks after enrolment. This will allow assessment of the natural history of this form of Crohn's disease and ensure that any changes in CDAI and QOL after capsule endoscopy are not merely a result of this natural history.

ELIGIBILITY:
Inclusion Criteria:

* Patient will be 10 years and older
* Patient suffers from abdominal pain and/or diarrhea for the last 6 weeks and/or expresses extra-intestinal manifestations of CD
* Patient has at least one of the following over the preceding 6 months (plus symptoms suspicious of small bowel Crohn's Disease):

  * Positive inflammatory marker (ESR, CRP, thrombocytosis, leucocytosis, fecal lactoferrin, fecal α-1 antitrypsin)
  * Unexplained anemia,
  * Recurrent fever,
  * Weight loss (at least 10% of normal body weight in adults),
  * Hypoalbuminaemia (<3.5 g/dL),
  * Gastro-intestinal bleeding,
  * Chronic perianal disease (fistula, fissure),
  * Abnormal white cell scan
  * Positive ASCA
  * First degree relative of a person suffering from IBD (only for subjects without known IBD),
* Patient underwent standard evaluation that includes colonoscopy and attempted ileoscopy and also SBFT within six months prior to enrollment, which were non-diagnostic. Blood tests should have been done within one month of enrolment.

  * Patient or legal guardian agrees to sign the Informed Consent Form

Exclusion Criteria:

* Patients with indeterminate colitis where the purpose is only to make a definitive diagnosis and where the inclusion criteria are not otherwise met
* Patient is known to suffer from intestinal obstruction (symptoms such as severe abdominal pain with accompanying nausea or vomiting)
* Definite stricture seen on SBFT
* Patient had suspected GI stricture, a Given® Patency capsule was administered and Patient did not pass the Patency capsule.
* Patient has a pacemaker or other implanted electro-medical device
* Patient has known history of small bowel Crohn's disease
* Patient on treatment for active IBD
* Patient with suspected celiac disease that has not been excluded
* Patient on non-steroidal anti-inflammatory drugs including Aspirin, (twice weekly or higher) during the 3 months preceding enrolment
* Patient is pregnant
* Patient has any condition, which precludes compliance with study and/or device instructions, such as swallowing problems
* Patient suffers from life threatening conditions
* Patient is currently participating in another clinical study that may directly or indirectly affect the results of this study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: clinics
Sampling Method: Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
• To evaluate the yield of capsule endoscopy for the diagnosis of small bowel Crohn's disease in symptomatic patients with non-diagnostic standard work-up. | end of study

SECONDARY OUTCOMES:
• To assess the clinical impact made by CE in patients with clinically suspected small bowel Crohn's disease | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Warwick Selby, MD, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia
Locations (8):
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Repatriation General Hospital, Daw Park, South Australia
  - Eastern Health, Box Hill, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Cabrini Medical Centre, Malvern, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gardiner Hospital, Nedlands, Western Australia